CLINICAL TRIAL: NCT05109689
Title: A Randomized Controlled Trial of ACT-P Versus T4C for Community Reentry: Differential Efficacy and Mechanisms of Change
Brief Title: A Randomized Controlled Trial of ACT-P Versus T4C for Community Reentry
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Amie Zarling, Associate Professor, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-569-00
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Criminal Behavior; Violence
Keywords: Cognitive behavior therapy; Community reentry; Recidivism
MeSH Terms: conditions — Criminal Behavior; Recidivism

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into either ACT-P or T4C, two group programs that will run simultaneously.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-P (Experimental): ACT-P is a cognitive behavioral program based on acceptance and commitment therapy, and it has been modified for use in the prison setting.
  Interventions: Behavioral: ACT-P
- T4C (Active Comparator): Thinking for Change (T4C) is an evidence-based cognitive behavioral program focused on changing criminal thinking.
  Interventions: Behavioral: T4C

INTERVENTIONS:
Behavioral: ACT-P — ACT-P consists of five modules. The Big Picture sessions are interwoven throughout the 24 sessions to introduce the main concepts of the curriculum, such as values identification and awareness of criminal behaviors. The Emotion Regulation and Cognitive Skills modules focus on awareness of internal experiences; learning new ways to respond to internal experiences; identifying and stepping back from problematic/criminal thoughts and beliefs; awareness of behaviors in service of values versus behaviors in service of control/avoidance; and identifying steps for behavior change. The Behavioral Skills module focuses on practicing prosocial behaviors, such as speaking and listening effectively and conflict resolution. Finally, the Barriers to Change module addresses environmental or life circumstances that can hinder successful behavior change (e.g., toxic masculinity, substance use, and parenting difficulties).
  Arms: ACT-P
Behavioral: T4C — T4C is an integrated cognitive behavioral change program authored by Drs. Jack Bush, Barry Glick, and Juliana Taymans under a cooperative agreement with the National Institute of Corrections (NIC). The program is based on the principle that thinking controls how people act, and that to change the way people act, they have to control their thinking. T4C systematically presents the concept that thoughts cause one's behavior, and offenders learn to identify their own thought patterns that lead to risky behavior, and then to replace those maladaptive thoughts with new ones. T4C incorporates research from cognitive restructuring theory, social skills development, and the learning and use of problem solving skills.
  Other Names: Thinking for a Change
  Arms: T4C

SUMMARY:
The purpose of the proposed study is to determine the efficacy of Acceptance and Commitment Therapy for prisons (ACT-P) and Thinking for a Change (T4C) as reentry programs in a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
The proposed study will focus on medium to high risk adult males, currently institutionalized and approaching release, who will be randomized to Acceptance and Commitment Therapy for prisons (ACT-P) or the Thinking for a Change (T4C) program. ACT-P is a cognitive behavioral treatment that targets acceptance and mindfulness processes to reduce criminal behavior, and has been adapted for the prison setting. T4C is a widely used and well-established traditional cognitive behavioral program that targets changing criminal thinking.

The first aim of the study is to test the relative efficacy of the ACT-P intervention, compared to T4C, on recidivism. Recidivism will be measured in 3 ways: rearrests, reconvictions, and reincarceration during the 3 years post-release. A secondary aim is to test the theory of change and the proposed mechanisms of ACT-P and T4C. By focusing on the mechanisms that account for program success, it will provide insight into the theory of change underlying each program. Based on the theories underlying each treatment, we hypothesize differences in mechanisms of action between the two treatments. Given the emphasis in T4C on cognitive change, we predict stronger mediation effects in T4C for reductions in antisocial/criminal thinking. In contrast, we hypothesize that increases in psychological flexibility would be stronger mediators for ACT-P than for T4C.

ELIGIBILITY:
Inclusion Criteria:

* deemed medium or high risk according to the Iowa Risk Revised
* eligible and appropriate for cognitive programming as determined by normal operating procedures

Exclusion Criteria:

* court-mandated to either program

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rearrests, convictions, and reincarcerations | 3 years post-release
  Criminal activity

CONTACTS AND LOCATIONS:
Locations (1):
- Fort Dodge Correctional Facility, Fort Dodge, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are undecided right now.